CLINICAL TRIAL: NCT02061488
Title: Prospective, Monocentric, Crossover Randomized Trial, to Assess a New Closed-loop Algorithm in Type 1 Diabetes (Saddle Point Model Predictive Control : SP-MPC)
Brief Title: Assessment of a New Closed-loop Algorithm in Type 1 Diabetes (Saddle Point Model Predictive Control : SP-MPC) (PPA)
Acronym: PPA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2013-A01604-41; 35RC13_8806_PPA (Other: Rennes University Hospital)
Record Dates: First submitted 2014-02-11; First posted 2014-02-12 (Estimated); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Type 1 Diabetes
Keywords: Artificial pancreas, closed loop glucose control, model predictive control
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- open-loop night (Active Comparator)
  Interventions: Other: open-loop night
- closed-loop night (Experimental)
  Interventions: Other: closed-loop night

INTERVENTIONS:
Other: open-loop night — During the open-loop night the patient is using his insulin pump as usual
  Arms: open-loop night
Other: closed-loop night — During the closed-loop night glucose values measured by the sensor are collected every 15 minutes. The data are entered into the SP-MPC controler that calculate the insulin dose to be delivered. A diabetologist validates the insulin dose before the infusion (manually bolus infusion)
  Arms: closed-loop night

SUMMARY:
The purpose of the study is to assess a new closed-loop algorithm in type 1 diabetes (Saddle Point Model Predictive Control : SP-MPC)

DETAILED DESCRIPTION:
Ten patients will be assessed during a closed-loop night and an open-loop night in random order.

The primary objective is to assess the ability of SP-MPC controler to maintain euglycemia and avoid hypoglycaemia during the night, compared to open loop in type 1 diabetic patients treated by insulin pump.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 1 diabetes (C peptide negative) :
* 18 to 70 year old,
* with type 1 diabetes for more than 3 years,
* treated by insulin pump for more than 3 months,
* with previous CGM holter allowing preliminary settting of some of the SP-MPC parameters
* able to provide written informed consent.

Exclusion Criteria:

* pregnancy or breastfeeding,
* severe non stabilized diabetic retinopathy,
* cardiovascular event in the previous 6 months,
* infectious diseases with recent fever,
* anemia (hemoglobin < 11g/l),
* HbA1c > 10%,
* Current or recent (less than 4 weeks) oral or injectable corticosteroid treatment,
* creatinine clearance <40ml/mn,
* chronic alcoholism (weekly consumption of alcohol > 280g for men and > 140g for women),
* adults legally protected (under judicial protection, guardianship, or supervision), persons deprived of their liberty

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-03; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Assessment of time spent in target range (glycemia between 70 and 145 mg/dl) and in hypoglycemia (glycemia <70 mg/dl), during the night (11 PM to 8 AM) | 6 weeks
  Assessment of the ability of SP-MPC controler to maintain euglycemia and avoid hypoglycaemia during the night, compared to open loop in type 1 diabetic patients treated by insulin pump

SECONDARY OUTCOMES:
Assessment of time spent above 70 mg/dl, between 70-145 or 145-180 mg/dl and above 180 mg/dl (interstitial glucose) in the late post prandial period (9 to 11 PM) and during the night (11 PM to 8 AM) | 6 weeks
  Assessment of hypoglycemia and hyperglycemia cases, average glycemic balance, glycemic variability, insulin doses
Assessment of hypoglycemia occurrence during the night | 6 weeks
Assessment of area under the curves (70-180mg/dl) during the night | 6 weeks
Assessment of Low Blood Glucose Index (LBGI), High Blood Glucose Index (HBGI) and CONGA Index | 6 weeks
Assessment of insulin doses delivered between 9 PM and 8 AM | 6 weeks
Assessment of number of controller propositions rejected for security reasons | 6 weeks
Assessment of glucose values during the night (glycemia and interstitial glucose values) | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Guilhem, Principal Investigator — Rennes University Hospital
Locations (1):
- Rennes University Hospital, Rennes, France

REFERENCES:
- [Result] Guilhem I, Penet M, Paillard A, Carpentier M, Esvant A, Lefebvre MA, Poirier JY. Manual Closed-Loop Insulin Delivery Using a Saddle Point Model Predictive Control Algorithm: Results of a Crossover Randomized Overnight Study. J Diabetes Sci Technol. 2017 Sep;11(5):1007-1014. doi: 10.1177/1932296817717503. Epub 2017 Jul 5. PMID 28677416